CLINICAL TRIAL: NCT02713828
Title: A Phase I/II Study of Glembatumumab Vedotin in Patients With gpNMB-Expressing, Advanced or Metastatic Squamous Cell Carcinoma of the Lung
Brief Title: Study of Glembatumumab Vedotin in gpNMB-Expressing, Advanced or Metastatic SCC of the Lung
Acronym: PrE0504
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company discontinued further development of study drug for this indication
Sponsor: PrECOG, LLC. (Other)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrE0504; CDX011-54 (Other: Celldex Therapeutics)
Record Dates: First submitted 2016-03-08; First posted 2016-03-21 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Squamous Cell Carcinoma of the Lung
Keywords: gpNMB-Expressing Squamous Cell Carcinoma of the Lung; Stage IIIb; Stage IV; Advanced Squamous Cell Cancer of the Lung; Metastatic Squamous Cell Cancer of the Lung; gpNMB-Expressing; Glembatumumab Vedotin
MeSH Terms: interventions — glembatumumab vedotin; CR011-vcMMAE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I: Glembatumumab Vedotin (Experimental): Glembatumumab vedotin once every three weeks (q3w) by 90-minute intravenous (IV) infusion, until disease progression or intolerance. The Dose-Limiting Toxicity (DLT) evaluation period for determination of the appropriateness of dose-escalation will be through the end of the second treatment cycle.
  Interventions: Drug: Phase I: Glembatumumab Vedotin
- Phase II: Glembatumumab Vedotin (Experimental): Glembatumumab vedotin once every three weeks (q3w) by 90-minute intravenous (IV) infusion, until disease progression or intolerance. The Maximum Tolerated Dose (MTD) determined in Phase I will be used in Phase II.
  Interventions: Drug: Phase II: Glembatumumab Vedotin

INTERVENTIONS:
Drug: Phase I: Glembatumumab Vedotin — Escalation Phase: Three to 6 patients will be enrolled in each dose cohort based on a standard Phase I dose escalation scheme. For the dose-escalation, the starting dose of glembatumumab vedotin will be 1.9 mg/kg q3w (Cohort 1). In the event of ≥ 2 DLTs, the dose will de-escalate to Cohort -1 (1.3 mg/kg).
  Dose escalation from Cohort 1 to Cohort 2 (2.2 mg/kg) may proceed if three patients in Cohort 1 complete the DLT observation period with 0 DLTs, or if six patients in Cohort 1 complete the DLT observation period with 0 or 1 DLTs.
  Other Names: CDX-011; CR011-vcMMAE
  Arms: Phase I: Glembatumumab Vedotin
Drug: Phase II: Glembatumumab Vedotin — In Stage 1, approximately 20 eligible, treated patients will be enrolled. If ≥ 2 patients achieve a tumor response (Partial Response [PR] or Complete Response [CR]), an additional 15 eligible, treated patients will be enrolled in Stage 2, for a maximum total of 35 eligible, treated patients.
  Other Names: CDX-011; CR011-vcMMAE
  Arms: Phase II: Glembatumumab Vedotin

SUMMARY:
Patients with advanced or metastatic, gpNMB-expressing Squamous Cell Carcinoma (SCC) of the lung who have failed a prior platinum-based chemotherapy regimen will receive glembatumumab vedotin.

Glembatumumab vedotin consists of an antibody (a type of human protein) attached to a drug called Monomethyl Auristatin E (MMAE) that can kill cancer cells. Glembatumumab vedotin is intended to work by specifically directing the drug to the cancer cell. It attaches to a molecule on the cancer cell called gpNMB, and then releases the MMAE inside the tumor cell, which in turn causes the cell to die.

The purpose of this study is to see whether glembatumumab vedotin is effective in treating people who have advanced or metastatic squamous cell lung cancer that contains gpNMB, to examine how the body handles the drug and the side effects associated with glembatumumab vedotin.

DETAILED DESCRIPTION:
Lung cancer is the most frequent cancer in the world, with annual cases worldwide currently estimated at one million and increasing to 10 million by the year 2025. In the United States, despite the declining incidence in white males in recent years, lung cancer is still the second most frequent cancer in both men (next to prostate) and women (next to breast cancer).

This is an open-label, single arm study of glembatumumab vedotin, a fully-human IgG2 monoclonal antibody. The activity of glembatumumab vedotin may be greatest in patients who overexpress the target, gpNMB.

This study will include a dose-escalation phase to determine the maximum safe and tolerated dose. This will be followed by a 2-stage Phase II expansion. During Phase II Stage 1, approximately 20 eligible, treated patients will be enrolled. If ≥ 2 patients achieve a tumor response [Partial Response (PR) or Complete Response (CR)]; an additional 15 eligible, treated patients will be enrolled in Stage 2, for a maximum total of 35 eligible, treated patients.

Glembatumumab vedotin will be administered once every 3 weeks, as a 90-minute intravenous (IV) infusion.

Patients will continue treatment until disease progression or intolerance. Tumor assessments will be performed every six (±1) weeks for six months, and every nine (±2) weeks thereafter, until progression.

A tumor tissue sample (i.e., obtained during a previous procedure or biopsy) will be sent to a central laboratory and tested for gpNMB. Research blood samples will also be required.

ELIGIBILITY:
Inclusion Criteria:

1. Read, understood, and provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization after the nature of the study has been fully explained and must be willing to comply with all study requirements and procedures.
2. Male or female patients with metastatic, histologically- or cytologically-confirmed unresectable Stage IIIB or IV non-small cell lung cancer (NSCLC) of squamous histology (Staging per American Joint Committee on Cancer [AJCC], Edition 7). Mixed histology adenosquamous NSCLC will also be permitted.
3. Experienced progression/recurrence of disease during or subsequent to the most recent anti-cancer regimen.
4. Any number of prior lines of systemic therapy may have been received for advanced (recurrent, locally advanced, or metastatic) SCC of the lung, but at least one must have been a platinum-based chemotherapy regimen. Platinum therapy may be given on-label or as part of a clinical trial.
5. Lung cancer confirmed to express gpNMB, as assessed by immunohistochemistry at a central lab (using expression in ≥ 5% of tumor epithelial cells as a cut-off for positivity). This can be tested on archived tissue if available, although preferred tumor specimen is a biopsy after the most recent therapy.
6. Age ≥ 18 years.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1.
8. Measurable disease by RECIST 1.1 criteria. Target lesions selected for tumor measurements should be those where surgical resection or radiation are not indicated or anticipated.
9. Resolution of all toxicities related to prior therapies to ≤ NCI-CTCAE Grade 1 severity, except for alopecia, vitiligo, or endocrinopathies on replacement therapy.
10. Adequate bone marrow function as assessed by absolute neutrophil count (ANC) ≥ 1500/mm3; hemoglobin ≥ 9.0 g/dL, and platelet count ≥ 100,000/mm3.
11. Adequate renal function as assessed by serum creatinine ≤ 2.0 mg/dL; or calculated or 24-hour urine creatinine clearance >40 mL/min.
12. Serum albumin ≥ 3 g/dL.
13. Adequate liver function as assessed by total bilirubin ≤ 1.5x upper limit of normal (ULN), and alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5x ULN (≤ 5.0x ULN in the case of liver metastases). Patients with known Gilbert's syndrome may be enrolled with total bilirubin ≤ 3.0 mg/dL.
14. Both male and female patients of childbearing potential enrolled in this trial must use adequate birth control measures during the course of the trial and for at least one month after discontinuing study drug.
15. Willing to provide blood samples for research purposes.

Exclusion Criteria:

1. Received glembatumumab vedotin (CR011-vcMMAE; CDX-011) or other MMAE-containing agents previously.
2. Chemotherapy within 21 days or at least 5 half-lives prior to the planned start of study treatment; radiation outside the thorax within 14 days prior to the planned start of study treatment or thoracic radiation; antibody based therapy or investigational therapy within 28 days prior to the planned start of study treatment.
3. Neuropathy >NCI-CTCAE Grade 1.
4. Subjects with a history of allergic reactions attributed to compounds of similar composition to dolastatin or auristatin. Compounds of similar composition include Auristatin PHE as an anti-fungal agent, Auristatin PE (TZT-1027, Soblidotin, NSC-654663) as an anti-tumor agent and Symplostatin 1 as an anti-tumor agent.
5. Known brain metastases, unless previously treated and patients are neurologically returned to baseline except for residual signs and symptoms related to Central Nervous System (CNS) treatment and CNS lesions are not progressive in size and number for 4 weeks.
6. Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension, and congestive heart failure related to primary cardiac disease, a history of a serious uncontrollable arrhythmia despite treatment, ischemic or severe valvular heart disease, or a myocardial infarction within 6 months prior to the trial entry.
7. Active systemic infection requiring treatment. Infection controlled by oral therapy will not be exclusionary.
8. Subjects on immunosuppressive medications such as azathioprine, mycophenolate mofetil, cyclosporine or require chronic corticosteroid use (defined as ≥ 3 months of prednisone dose equivalent of ≥ 10 mg).
9. The MMAE component of glembatumumab vedotin is primarily metabolized by CYP3A. Patients taking strong CYP3A inhibitor and inducers are excluded in Phase I (the dose escalation portion), to minimize the effect of these modulators on exposure, tolerability and dose selection.
10. History of other malignancy except for adequately treated basal or squamous cell skin cancer, curatively treated in situ disease, or any other cancer from which the patient has been disease-free for ≥ 2 years.
11. Pregnant or breast-feeding women.
12. Subjects must not be on home oxygen therapy (intermittent or continuous).
13. Any underlying medical condition that, in the Investigator's opinion, will make the administration of study treatment hazardous to the patient, or would obscure the interpretation of adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04-10 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rathi Pillai, MD, Study Chair — PrECOG, LLC.
Locations (10):
- United States (10):
  - University of Miami Hospital, Miami, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Ochsner Medical Center, New Orleans, Louisiana
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Stony Brook University, Stony Brook, New York
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - West Virginia University, Morgantown, West Virginia
  - Gundersen Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Glembatumumab Vedotin: Glembatumumab vedotin once every three weeks (q3w) by 90-minute intravenous (IV) infusion, until disease progression or intolerance. The Dose-Limiting Toxicity (DLT) evaluation period for determination of the appropriateness of dose-escalation will be through the end of the second treatment cycle.
  Phase I: Glembatumumab Vedotin: Escalation Phase: Three to 6 patients will be enrolled in each dose cohort based on a standard Phase I dose escalation scheme. For the dose-escalation, the starting dose of glembatumumab vedotin will be 1.9 mg/kg q3w (Cohort 1). In the event of ≥ 2 DLTs, the dose will de-escalate to Cohort -1 (1.3 mg/kg).
  Dose escalation from Cohort 1 to Cohort 2 (2.2 mg/kg) may proceed if three patients in Cohort 1 complete the DLT observation period with 0 DLTs, or if six patients in Cohort 1 complete the DLT observation period with 0 or 1 DLTs.
Period: Overall Study
Arm/Group | Phase I: Glembatumumab Vedotin | Phase II: Glembatumumab Vedotin
Started | 13 | 0
Completed | 8 | 0
Not Completed | 5 | 0
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — study terminated but patient allowed to | 2 | 0

BASELINE CHARACTERISTICS:
Population: The study terminated early during the phase I portion of the trial
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Glembatumumab Vedotin | Phase II: Glembatumumab Vedotin | Total
Number analyzed (Participants) | 13 | 0 | 13
Age, Continuous [Median (Full Range); unit: years] | 63 [52 to 75] |  | 63 [52 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 |  | 6
  Male | 7 |  | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 11 |  | 11
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
ECOG Performance Status [Count of Participants; unit: Participants] — PS 0: Fully active, able to carry on all pre-disease performance without restriction; PS 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature e.g. light house work, office work.
  Participants
    PS 0 | 2 |  | 2
    PS 1 | 11 |  | 11
Prior lines of treatment [Count of Participants; unit: Participants]
  1 | 5 |  | 5
  2 | 4 |  | 4
  >=3 | 3 |  | 3
  unknown | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Determine Maximum Tolerated Dose (MTD)
Description: To determine the Maximum Tolerated Dose (MTD) by number of participants with DLTs.
Time Frame: 42 (±3) days
Measure: Number; unit: mg/kg
Arm/Group | Phase I: Glembatumumab Vedotin
Number analyzed (Participants) | 13
mg/kg | NA — PrECOG received notification from Celldex noting the suspension of glembatumumab vedotin development and the closure of the PrE0504 study before the MTD was determined and the phase I part of the study was completed.

2. Primary Outcome: Phase II: Objective Response Rate (ORR)
Description: Determine the anti-tumor activity, as assessed by ORR in accordance with RECIST 1.1, of the MTD of glembatumumab vedotin in patients with advanced gpNMB-expressing SCC of the lung.
Time Frame: 40 months
Population: The study terminated early during the phase I portion of the trial
Arm/Group | Phase II: Glembatumumab Vedotin
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0.
Description: To further characterize the safety of glembatumumab vedotin by the number of participants with abnormal laboratory values and/or adverse events related to treatment (including Serious Adverse Events and Other Adverse Events).
Time Frame: 23 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Glembatumumab Vedotin
Number analyzed (Participants) | 13
Participants | 13

4. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR assessed in accordance with RECIST 1.1.
Time Frame: 23 months
Population: 1 patient achieved partial response. The duration of this patient's response is at least 9.4 months, with response ongoing at the time of final report.
Measure: Number; unit: months
Arm/Group | Phase I: Glembatumumab Vedotin
Number analyzed (Participants) | 1
months | 9.4

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS assessed in accordance with RECIST 1.1.
Time Frame: 23 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I: Glembatumumab Vedotin
Number analyzed (Participants) | 13
months | 2.5 [1.6 to NA] — Upper limit can't be estimated.

6. Secondary Outcome: Overall Survival (OS)
Description: OS assessed in accordance with RECIST 1.1.
Time Frame: 23 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I: Glembatumumab Vedotin
Number analyzed (Participants) | 13
months | 5.8 [2.5 to NA] — Upper limit can't be estimated

ADVERSE EVENTS:
Time Frame: 23 months
Arm/Group | Phase I: Glembatumumab Vedotin
All-Cause Mortality (participants affected / at risk) | 7/13
Serious Adverse Events (participants affected / at risk) | 9/13
Other Adverse Events (participants affected / at risk) | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Glembatumumab Vedotin (N=13)
Abdominal pain (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Glembatumumab Vedotin (N=13)
Abdominal pain (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Metabolism and nutrition disorders Dehydration (Metabolism and nutrition disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Candida infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Eye pain (Eye disorders) | 1
Fatigue (General disorders) | 3
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Iridocyclitis (Eye disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Malaise (General disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT02713828/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT02713828/SAP_001.pdf